CLINICAL TRIAL: NCT02124499
Title: Genetic Variants and Perioperative Morbidity and Mortality
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 041/09
Record Dates: First submitted 2014-04-04; First posted 2014-04-28 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Analgesia; Surgical Procedure, Operative
Keywords: anesthesia recovery period; postoperative complications; pain; pain measurement; postoperative nausea and vomiting; quality of life; genetic association study
MeSH Terms: conditions — Agnosia; Postoperative Complications; Pain; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (plasma and cells) or mucosal swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All patients: Patients undergoing elective surgery with anesthesia

SUMMARY:
Prospective association study to analyse perioperative patients' outcome. Outcome comprises intraoperative and postoperative complications e.g. cardio-vascular events, allergic reactions, Possible variables which might have on influence: patient- and surgery-related data, patients' genetic background etc.

DETAILED DESCRIPTION:
Background Anesthesia and surgery are related to unwanted adverse events, side effects and postoperative discomfort. Whereas severe complications like cardiovascular events are rare, postoperative side effects like nausea and vomiting, pain, long-lasting pain and pain related interference of daily activities are frequent. The question arises which patient is at specific risk for this sequelae. Pre-exiting predisposing factors (e.g. patients' genetic background), surgery and anesthesia related variables (drugs, techniques administered for anesthesia and analgesia) as well as psychological and social factors might influence the outcome.

In this prospective association study these variables will be investigated in a well-described patient cohort presenting for elective surgery.

Objective

The aim of this study is to associate perioperative and postoperative complications and side effects as well as long-term outcome after surgery to patient- and surgery-related variables, including genetic variants.

Methods

Prospective association study performed in two independent patient cohorts.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Written informed consent
* Scheduled surgery

Exclusion Criteria

* No informed consent
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2011-01-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | Up to 48 hours after surgery
  Percent of patients with no PONV, medium PONV and severe PONV PONV outcome measured by a composite score: number of episodes of vomiting + severity of nausea (NRS score) + need for antiemetic treatment Patients with no PONV are compared to those with intermediate and severe PONV

SECONDARY OUTCOMES:
Pain related impairment after surgery | up to 2 days after surgery
  Measured by the International Pain Outcomes Questionnaire
Pain related impairment of patients with chronic pain after surgery versus patients without chronic pain after surgery | up to one year after surgery
  Measured by the Brief Pain Inventory (BPI)
Cardio-vascular events after surgery | Up to 30 days after surgery
  Measured by a score for major adverse cardiac events (MACE)
Pain related impairment of patients with chronic neuropathic pain (DN4 positive) after surgery versus patients without neuropathic pain after surgery | up to one year after surgery
  Measured by the Brief Pain Inventory (BPI)
What influences pain related impairment after bariatric surgery | up to 1 year after surgery
  Measurement of patient reported outcome by the BPI (Brief Pain Inventory).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Stüber, Prof. MD, Study Chair — Department of Anaestheisolpogy + Pain Medicine, Inselspital, University of Bern; Ulrike M Stamer, MD, Principal Investigator — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern, Bern, Switzerland